CLINICAL TRIAL: NCT03992781
Title: NON-INTERVENTIONAL STUDY TO REVIEW THE CHANGES OF DEPRESSION AFTER FIRST-YEAR OF TOFACITINIB TREATMENT IN RHEUMATOID ARTHRITIS (XELJANZ (Registered))
Brief Title: Changes of Depression After First-year of Tofacitinib in RA Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921330; NCT03992781 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2019-05-24; First posted 2019-06-20 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Newly prescribed tofacitinib: patients who were newly prescribed tofacitinib at baseline and who scored at least 11 points on CUDOS scale

SUMMARY:
12-month, single arm, prospective, non-interventional, multi-center study according to Czech legal definitions (Law 378/2007 Sb.).The primary objective of this study is to describe and evaluate the changes of depression level within 12 months from the start of tofacitinib therapy in patients with RA and at least minimal level of depression. Primary goal is to find out if treatment by tofacitinib reduces the depression by at least 10% during 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years.
* Moderate to severe activity of rheumatoid arthritis (DAS28 ≥3.2).
* Patient for whom the physician decision has been made to initiate a treatment with Tofacitinib.
* Patient with at least minimal level of depression (CUDOS questionnaire ≥11 points).
* Capable of understanding and signing a written informed consent form.
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study is a requirement for inclusion into this study.

Exclusion Criteria:

* Patients unwilling/unable to fill in printed patient questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who are initiated on tofacitinib as part of a usual care setting.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Czechia (6):
  - Thomayerova nemocnice, Prague, Czech Republic
  - Revmatologie s.r.o., Brno
  - Rheuma s.r.o., Břeclav
  - Artroscan, s.r.o., Ostrava - Trebovice
  - Revmatologicky ustav, Prague
  - Revmatologicke centrum s.r.o., Velké Bílovice

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921330

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were diagnosed with moderate to severe rheumatoid arthritis (RA), initiated tofacitinib treatment for the first time and scored at least 11 points on clinically useful depression outcome scale (CUDOS) were enrolled. Participants were followed up for 12 months.
Groups:
- All Participants: All eligible participants who initiated tofacitinib treatment at Visit 1 (Day 1) in real world setting per routine care and in accordance with local marketing authorization, were included in this observational study.
Period: Overall Study
Arm/Group | All Participants
Started | 73
Safety Analysis Set | 70
Full Analysis Set | 62
Completed | 62
Not Completed | 11
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least one dose of tofacitinib.
Arm/Group | All Participants
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: CUDOS Score: Baseline (Visit 1) and 12 Months (Visit 3)
Description: The CUDOS questionnaire assessed the level of depression in the past week. It consisted of 18 questions. For each question the participant indicated how well it described his/her feelings during past week on the following scale: 0 = not at all true, 1 = rarely true, 2 = sometimes true, 3 = often true and 4 = almost always true. The result of this questionnaire was the sum of responses to all questions and therefore the overall possible CUDOS score ranged from 0 to 72, higher score indicated more severe depression. Absolute values of CUDOS score at baseline (Visit 1) and 12 Months (Visit 3) are reported in descriptive data below. Mean relative change was calculated by averaging the relative changes of each of the participants (sum of all relative changes divided by the number of participants) and was reported in the statistical section.
Time Frame: Baseline (Visit 1), 12 Months (Visit 3)
Population: Full analysis set (FAS) included all participants who received at least one dose of tofacitinib and had the data for evaluation of primary hypothesis, which means CUDOS reported both at baseline and visit 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 62
Units on a scale
  Baseline (Visit 1) | 21.97 (9.45)
  12 Months (Visit 3) | 9.29 (6.71)
Statistical Analysis 1: Comparison: All Participants; Relative change in CUDOS score between Visit 3 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -53.1

2. Secondary Outcome: CUDOS Score: Baseline (Visit 1) and 6 Months (Visit 2)
Description: The CUDOS questionnaire assessed the level of depression in the past week. It consisted of 18 questions. For each question the participant indicated how well it described his/her feelings during past week on the following scale: 0 = not at all true, 1 = rarely true, 2 = sometimes true, 3 = often true and 4 = almost always true. The result of this questionnaire was the sum of responses to all questions and therefore the overall possible CUDOS score ranged from 0 to 72, higher score indicated more severe depression. Absolute values of CUDOS score at baseline (Visit 1) and 6 Months (Visit 2) are reported in descriptive data below. Mean relative change was calculated by averaging the relative changes of each of the participants (sum of all relative changes divided by the number of participants) and was reported in the statistical section.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2)
Population: FAS included all participants who received at least one dose of tofacitinib and had the data for evaluation of primary hypothesis, which means CUDOS reported both at baseline and visit 3.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 62
Units on a scale
  Baseline (Visit 1) | 21.97 (9.45)
  6 Months (Visit 2) | 12.79 (8.71)
Statistical Analysis 1: Comparison: All Participants; Relative change in CUDOS score between Visit 2 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -35.4

3. Secondary Outcome: CUXOS Score: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Description: The clinically useful anxiety outcome scale (CUXOS) questionnaire assessed the level of anxiety in the past week. It consisted of 20 questions. For each question the participant indicated how well it described his/her feelings during past week on the following scale: 0 = not at all true, 1 = rarely true, 2 = sometimes true, 3 = often true and 4 = almost always true. The result of this questionnaire was the sum of responses to all questions and therefore the overall possible CUXOS score ranged from 0 to 80, higher score indicated higher anxiety level. Absolute values of CUXOS score at baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3) are reported in descriptive data below. Mean relative change was calculated by averaging the relative changes of each of the participants (sum of all relative changes divided by the number of participants) and was reported in the statistical section.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 62
Units on a scale
  Baseline (Visit 1) | 20.45 (14.21)
  6 Months (Visit 2) | 12.24 (11.31)
  12 Months (Visit 3) | 8.21 (8.66)
Statistical Analysis 1: Comparison: All Participants; Relative change in CUXOS score between Visit 2 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -33.2
Statistical Analysis 2: Comparison: All Participants; Relative change in CUXOS score between Visit 3 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -47.1

4. Secondary Outcome: JSEQ Score: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Description: The Jenkins sleep evaluation questionnaire (JSEQ) questionnaire assessed the level of insomnia, sleep disturbance in the past month. It consisted of 4 questions related to 1) trouble falling asleep, 2) trouble staying asleep, 3) waking up several times per night, and 4) waking up feeling tired and worn out after a usual amount of sleep. The response alternatives were: 0 = not at all, 1 = 1-3 days, 2 = 4-7 days, 3 = 8-14 days, 4 = 15-21 days, and 5 = 22-30 days. The result of this questionnaire was the sum of responses to all questions and therefore the overall possible JSEQ score ranged from 0 to 20, higher score indicated lower sleep quality. Absolute values of JSEQ score at baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3) are reported in descriptive data below. Mean relative change was calculated by averaging the relative changes of each of the participants (sum of all relative changes divided by the number of participants) and was reported in the statistical section.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 62
Units on a scale
  Baseline (Visit 1) | 9.40 (4.78)
  6 Months (Visit 2) | 6.63 (4.61)
  12 Months (Visit 3) | 5.48 (3.52)
Statistical Analysis 1: Comparison: All Participants; Relative change in JSEQ score between Visit 2 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -27.6
Statistical Analysis 2: Comparison: All Participants; Relative change in JSEQ score between Visit 3 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -34.5

5. Secondary Outcome: VAS Score: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Description: Participants assessed how much arthritis impacted their life using a 100 millimeter (mm) visual analogue score (VAS) by placing a mark on the scale between 0 (not affecting) and 100 (maximal impact), which corresponded to the level arthritis affected their life. The score ranged from 0 mm to 100 mm, higher score indicated higher impact of arthritis on participants life. Absolute values of VAS score at baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3) are reported in descriptive data below. Mean relative change was calculated by averaging the relative changes of each of the participants (sum of all relative changes divided by the number of participants) and was reported in the statistical section.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: FAS included all participants who received at least one dose of tofacitinib and had the data for evaluation of primary hypothesis, which means CUDOS reported both at baseline and visit 3. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 38
Units on a scale
  Baseline (Visit 1) | 61.42 (18.62)
  6 Months (Visit 2) | 33.58 (20.34)
  12 Months (Visit 3) | 33.75 (26.57)
Statistical Analysis 1: Comparison: All Participants; Relative change in VAS score between Visit 2 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -43.4
Statistical Analysis 2: Comparison: All Participants; Relative change in VAS score between Visit 3 and Visit 1 was tested by ratio t-test (paired t-test of logarithm) at 0.05 alpha level. This was expressed in percentage; Test type: Superiority; p < 0.001, t-test; Relative change = -35.4

6. Secondary Outcome: Number of Participants Who Took at Least 1 Concomitant Treatment of Mental Illness Per Study Visit
Description: Number of participants who took at least 1 concomitant treatment like antidepressants, anxiolytics and hypnotics were reported in this outcome measure. Participants could have been counted in more than one category.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 62
Participants
  Visit 1: Antidepressants | 4
  Visit 1: Anxiolytics | 1
  Visit 1: Hypnotics | 5
  Visit 2: Antidepressants | 2
  Visit 2: Anxiolytics | 0
  Visit 2: Hypnotics | 3
  Visit 3: Antidepressants | 5
  Visit 3: Anxiolytics | 0
  Visit 3: Hypnotics | 2

7. Secondary Outcome: Number of Participants With Change in Dosage of Concomitant Medication Between 12 Months (Visit 3) and Baseline (Visit 1)
Description: Number of participants with change in number of used medications and in their dosage between 12 Months (Visit 3) and Baseline (Visit 1) were reported in this outcome measure.
Time Frame: Baseline (Visit 1), 12 Months (Visit 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 62
Participants
  Antidepressants | 1
  Anxiolytics | 1
  Hypnotics | 3

8. Secondary Outcome: Absolute Change From Baseline in DAS28-4 (CRP) at 6 Months (Visit 2) and 12 Months (Visit 3)
Description: Disease activity score 28-4 (DAS28-4) C-reactive protein (CRP) was calculated from 28-tender joint counts and 28-swollen joint counts, CRP (milligram per liter [mg/L]) and patient global assessment (PGA); participant assessed overall disease activity on VAS, score: 0 [no arthritis] to 100 [extreme arthritis]. DAS 28 -4 CRP = 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.36*In (CRP in mg/1 + 1) + 0.014*PtGA + 0.96; ln = natural logarithm, sqrt = square root of, mg = milligram, PtGA = patient's global assessment of health. DAS28-4 (CRP) lower than (<) 2.6 = RA in remission, 2.6 to 3.2 = low level of disease activity, 3.2 to 5.1 = active disease, may require change of treatment and greater than (>) 5.1 = very active disease, required careful monitoring and change of treatment. Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 62
Units on a scale
  Absolute change at Visit 2 | -3.01 (1.19)
  Absolute change at Visit 3 | -3.06 (1.41)

9. Secondary Outcome: Number of Participants Achieving Remission as Assessed by DAS28-4 (CRP) < 2.6
Description: Remission was defined as DAS28-4 (CRP) < 2.6. DAS28-4 CRP was calculated from 28-tender joint counts and 28-swollen joint counts, CRP (mg/L) and PGA; participant assessed overall disease activity on VAS, score: 0 [no arthritis] to 100 [extreme arthritis]. DAS 28 -4 CRP = 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.36*In (CRP in mg/1 + 1) + 0.014*PtGA + 0.96; ln = natural logarithm, sqrt = square root of, mg = milligram, PtGA = patient's global assessment of health. DAS28-4 (CRP) < 2.6 = RA in remission, 2.6 to 3.2 = low level of disease activity, 3.2 to 5.1 = active disease, may require change of treatment and > 5.1 = very active disease, required careful monitoring and change of treatment. Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 62
Participants
  Visit 1 | 0
  Visit 2 | 27
  Visit 3 | 26

10. Secondary Outcome: Number of Participants Achieving LDA as Assessed by DAS28-4 (CRP) < 3.2
Description: Low disease activity (LDA) was defined as DAS28-4 (CRP) < 3.2. DAS28-4 CRP was calculated from 28-tender joint counts and 28-swollen joint counts, CRP (mg/L) and PGA; participant assessed overall disease activity on VAS, score: 0 [no arthritis] to 100 [extreme arthritis]. DAS 28 -4 CRP = 0.56*sqrt (TJC28) + 0.28*sqrt (SJC28) + 0.36*In (CRP in mg/1 + 1) + 0.014*PtGA + 0.96; ln = natural logarithm, sqrt = square root of, mg = milligram, PtGA = patient's global assessment of health. DAS28-4 (CRP) < 2.6 = RA in remission, 2.6 to 3.2 = low level of disease activity, 3.2 to 5.1 = active disease, may require change of treatment and > 5.1 = very active disease, required careful monitoring and change of treatment. Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 62
Participants
  Visit 1 | 0
  Visit 2 | 40
  Visit 3 | 44

11. Secondary Outcome: Change From Baseline in EuroQol Five Dimension - 3 Level (EQ-5D-3L) Health State Profile at 6 Months (Visit 2) and 12 Months (Visit 3)
Description: EQ-5D-3L designed to assess impact on health-related quality of life in 5 domains: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each domain had 3 responses and scored from 1-3 (1=no problems; 2=some problems; 3=extreme problems). The mean of the summed score ranged from 1 to 3 with "1" corresponding to no problems and "3" corresponding to severe problems, where higher score indicated more severe problems. The EQ-5D-3L index score summarized each possible health state on a numerical scale ranging from -0.594 to 1. A score of 1 indicated full health, score of 0 indicated a state equivalent to being dead, and score lower than 0 indicated a state equivalent to the worst possible health status. Higher score indicated a better quality of life.
Time Frame: Baseline (Visit 1), 6 Months (Visit 2) and 12 Months (Visit 3)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 62
Units on a scale
  Change at Visit 2 | 0.157 (0.231)
  Change at Visit 3 | 0.179 (0.271)

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant who received study intervention without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and all non-SAEs. TEAEs were defined as newly occurring (not present at baseline) or worsening after first dose of study treatment.
Time Frame: From start of study treatment to 12 months post treatment initiation
Population: The safety analysis set included all participants who received at least one dose of tofacitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 70
Participants | 15

ADVERSE EVENTS:
Time Frame: From start of study treatment to 12 months post treatment initiation
Description: Same event may appear as both non-SAE and SAE but what is presented are distinct events. Event may be categorized as serious in 1 participant and non-serious in other, or participant may have experienced both serious and non-serious event. Safety population included all participants who received at least 1 dose of tofacitinib.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 1/70
Other Adverse Events (participants affected / at risk) | 15/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=70)
Thrombopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=70)
Thrombopenia (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Dryness of eyes (Eye disorders) | 1
Dryness oral (Gastrointestinal disorders) | 1
Drug effect lack of (General disorders) | 5
Acute bronchitis (Infections and infestations) | 1
Cold (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 1
Post herpetic neuralgia (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Virosis (Infections and infestations) | 2
Hematuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT03992781/Prot_SAP_000.pdf